CLINICAL TRIAL: NCT03552159
Title: Behavioral Activation for Dementia Caregivers: Scheduling Pleasant Events and Enhancing Communications
Brief Title: Behavioral Activation for Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other); Stanford University (Other); United Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCPF2012
Record Dates: First submitted 2018-05-30; First posted 2018-06-11 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2018-05

CONDITIONS: Dementia Caregivers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation (Experimental): For the first 4 weeks,participants received psychoeducation about the symptoms and associated behavioral changes of dementia and the possible effects on the caregivers, t the physical, social and psychological consequences of stress, event scheduling and communication skills. After psychoeducation, eight bi-weekly behavioral activation sessions were administered, focusing pleasant event scheduling and effective communications.
  Interventions: Behavioral: Behavioral activation; Other: Psychoeducation
- Psychoeducation (Active Comparator): For the first 4 weeks, participants were taught about the symptoms and associated behavioral changes of dementia and the possible effects on the caregivers, the physical, social and psychological consequences of stress, event scheduling and communication skills. After psychoeducation, eight biweekly phone sessions of general support but not behavioral activation.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: Behavioral activation — Activity scheduling, monitoring, review and re-scheduling
  Arms: Behavioral Activation
Other: Psychoeducation — Education on dementia, caregiving stress, event scheduling and communication skills

SUMMARY:
This project was designed to test a model targeted intervention for dementia caregivers telephone program consisting of both psychoeducation and behavioral activation components to reduce the burden of caregivers. The program is delivered by telephone to increase accessibility and sustainability for caregivers.

DETAILED DESCRIPTION:
The study compared two telephone interventions using a four-month longitudinal randomized controlled trial. For the first four weeks, all participants received the same psychoeducation program via telephone. Then for the following four months, eight biweekly telephone follow-up calls were carried out. For these eight follow-up calls, participants were randomized into either one of the two following groups with different conditions. For the Psychoeducation with BA (PsyED-BA) group, participants would receive eight biweekly sessions of BA practice focused on pleasant event scheduling and improving communications. For the Psychoeducation only (PsyED Only) group, there would be eight biweekly sessions of general discussion of psychoeducation and related information

ELIGIBILITY:
Inclusion Criteria:

They were caregivers aged 25 or above and must have be caring for a care recipient diagnosed with Alzheimer's disease for at least 3 months. They should be the primary caregiver and a spouse, kin (e.g. daughter/son or daughter/son-in-law) or sibling of the care recipient.

Exclusion Criteria:

To ensure intervention fidelity, participants who showed signs of severe intellectual deficits, demonstrate suicidal ideation, exhibit evidence of psychotic disorders, or cannot read or speak fluent Chinese / Cantonese were excluded.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms | Change from baseline through study completion, an average of about 5 months
  Measured by CES-D

SECONDARY OUTCOMES:
Sense of Burden | Change from baseline through study completion, an average of about 5 months
  Measured by Zarit Burden Scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Fraile E, Ballesteros J, Rueda JR, Santos-Zorrozua B, Sola I, McCleery J. Remotely delivered information, training and support for informal caregivers of people with dementia. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD006440. doi: 10.1002/14651858.CD006440.pub3. PMID 33417236
- [Derived] Au A, Yip HM, Lai S, Ngai S, Cheng ST, Losada A, Thompson L, Gallagher-Thompson D. Telephone-based behavioral activation intervention for dementia family caregivers: Outcomes and mediation effect of a randomized controlled trial. Patient Educ Couns. 2019 Nov;102(11):2049-2059. doi: 10.1016/j.pec.2019.06.009. Epub 2019 Jun 26. PMID 31279613